CLINICAL TRIAL: NCT06605326
Title: Subcutaneous Treprostinil as a Bridge to Lung Transplantation in Severe Pulmonary Hypertension: A Single-Arm Retrospective Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhibin Xu, Principal Investigator, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022K-48
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Chronic Lung Disease-Associated Pulmonary Hypertension; Lung Transplantation; Heart Failure
Keywords: Subcutaneous Treprostinil; NYHA Functional Class; 6-Minute Walk Distance; Primary Graft Dysfunction (PGD); Retrospective Study; Single-Arm Study
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Heart Failure; Primary Graft Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a single-arm, retrospective study in which all enrolled patients received subcutaneous treprostinil as a bridge therapy for lung transplantation. The study evaluates the efficacy and safety of the treatment in patients with severe pulmonary hypertension, including both PAH and CLD-PH. No randomization or control group is included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subcutaneous Treprostinil Group (Experimental): Patients in this group received subcutaneous treprostinil, starting at a dose of 1.25 to 4 ng/kg/min and gradually titrated according to patient response. The target dose was over 20 ng/kg/min after 3 months of treatment. All patients were referred for lung transplantation during or after treprostinil treatment.
  Interventions: Drug: Subcutaneous Treprostinil

INTERVENTIONS:
Drug: Subcutaneous Treprostinil — Patients in this group received subcutaneous treprostinil, starting at a dose of 1.25 to 4 ng/kg/min and gradually titrated according to patient response. The target dose was over 20 ng/kg/min after 3 months of treatment. All patients were referred for lung transplantation during or after treprostinil treatment.

SUMMARY:
This single-arm, retrospective study aims to evaluate the safety and efficacy of subcutaneous treprostinil as a bridge therapy for lung transplantation in patients with severe pulmonary hypertension (PH). A total of 46 patients with either pulmonary arterial hypertension (PAH) or chronic lung disease-associated PH (CLD-PH) were included, all of whom were referred for lung transplantation between January 1, 2015, and September 1, 2024. The study examines changes in clinical, functional, and hemodynamic parameters following 3-6 months of treprostinil therapy.

DETAILED DESCRIPTION:
This study evaluates the use of subcutaneous treprostinil as a bridge therapy for lung transplantation in patients with severe pulmonary hypertension (PH), including both pulmonary arterial hypertension (PAH) and chronic lung disease-associated PH (CLD-PH). This retrospective, single-center study included 46 patients treated between January 1, 2015, and September 1, 2024. All patients experienced significant clinical and hemodynamic impairment at the time of treprostinil initiation. The primary aim was to assess improvements in NYHA functional class and 6-minute walk distance (6-MWD) following 3-6 months of therapy. Secondary outcomes included NT-proBNP levels, echocardiographic parameters, and post-transplantation survival rates. The study also analyzed the incidence of primary graft dysfunction (PGD) and the continued use of treprostinil post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe pulmonary hypertension (PAH or CLD-PH) requiring lung transplantation
* Age 18 years or older
* Able to provide informed consent

Exclusion Criteria:

* Patients with PH caused by left heart disease
* Patients unable to undergo lung transplantation due to medical conditions
* Patients with a history of severe drug allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in NYHA Functional Class | Baseline to 3-6 months after treatment initiation
  The change in NYHA functional class will be assessed after 3-6 months of treatment with subcutaneous treprostinil. Improvement will be defined as a reduction in class (e.g., from class IV to class III or II).
Improvement in 6-Minute Walk Distance (6-MWD) | Baseline to 3-6 months after treatment initiation
  The 6-minute walk distance (6-MWD) will be measured at baseline and after 3-6 months of subcutaneous treprostinil treatment to evaluate the improvement in exercise capacity.

SECONDARY OUTCOMES:
Change in NT-proBNP Levels | Baseline to 3-6 months after treatment initiation
  NT-proBNP levels will be measured before and after treatment to assess changes in cardiac function.

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) from this study. Due to privacy concerns and the sensitive nature of the health data collected, the research team has decided not to make individual-level data available to external researchers. All data will remain confidential and will be used solely for the purposes of this study, in compliance with institutional and ethical guidelines.